CLINICAL TRIAL: NCT00144274
Title: Efficacy and Tolerability of Ambroxol Lozenges 20mg in Relieving the Pain of Sore Throat in Adolescent Patients With Acute Viral Pharyngitis - A Randomised, Double-blind, Placebo-controlled Parallel Group Study. AMBROSIA: Ambroxol Lozenges In Sore Throat In Adolescents
Brief Title: Ambroxol Lozenges 20mg in Relieving the Pain of Sore Throat in Adolescent Patients With Acute Viral Pharyngitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18.487
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis

INTERVENTIONS:
Drug: Ambroxol Lozenge

SUMMARY:
The purpose of this trial is to investigate efficacy and tolerability of lozenges containing 20mg am broxol hydrochloride relative to placebo in relieving pain of sore throat in adolescent patients suf fering from acute viral pharyngitis. The primary endpoint is the time-weighted average of the pain intensity difference from pre-dose bas eline over the first 3 hours after the first lozenge expressed as a ratio of the pre-dose baseline ( SPIDnorm).

DETAILED DESCRIPTION:
The purpose of this trial is to investigate efficacy and tolerability of lozenges containing 20mg am broxol hydrochloride relative to placebo in relieving pain of sore throat in adolescent patients suf fering from acute viral pharyngitis. The pain intensity will be assessed by the patient on a 6-point rating scale before taking the first lozenge and 30, 60, 120 and 180 minutes thereafter. The patient enters the rating in the patient's diary.

Study Hypothesis:

It will be tested whether a statistically significant difference exists in the S PIDnorm after the intake of the 1st lozenge between the group treated with ambro xol lozenges and the group treated with placebo lozenges.

Comparison(s):

Placebo comparison

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients having a sore throat with acute viral pharyngitis.
2. Female and male patients from 12 and less than 18 years of age.
3. The throat pain intensity is rated at least "moderate" on the VRS(PI).
4. Written Informed Consent is given by the patient's parent/legal guardian, an d the patient is able to give Assent.
5. Compliance by the patient seems guaranteed, and the patient seems to be able to understand and complete the patient diary.
6. Patient able to remain at the doctor's practice for the initial 3 hours follo wing the first intake of study medication, or known reliable patient, and able t o return for the study visits.

EXCLUSION CRITERIA

1. Female patients who have begun menstruating and are:

   1. Pregnant
   2. Currently breastfeeding
   3. Of child-bearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the study. Acceptable methods of birth control include surgical sterilisation, intra uterine device, oral, implantable or injectable contraceptives. Abstinenc e can be used as contraception, at the discretion of the investigator.
2. Patients with symptoms of primarily bacterial pharyngitis or bacterial secon dary infection (clinical findings inter alia assessment of exudate).
3. First indication of symptoms of acute pharyngitis (e.g. sore throat) occurre d more than 3 days ago.
4. Patients who suffered from acute viral or bacterial pharyngitis in the past 4 weeks.
5. Patient who in the past week, or during the study will require treatment with the following: antibiotics analgesics anti-inflammatory agents steroids fo r oral, inhaling or topical application expectorants or antitussives. No phys ical therapy (e.g. throat compress) may be applied during the trial.
6. Patients with mouth breathing as a result of nasal congestion.
7. Known hypersensitivity to Ambroxol or to auxiliary substances contained in t he lozenge.
8. Previous and/or existing tumour condition.
9. Alcohol, and/or drug abuse.
10. Any clinical condition which, in the opinion of the investigator would not a llow safe completion of the protocol and safe administration of trial medication.
11. Any investigational therapy within 30 days prior to randomisation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220
Dates: Start 2005-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11

PRIMARY OUTCOMES:
The primary endpoint is the time-weighted average of the pain intensity difference from pre-dose baseline over the first 3 hours after the first lozenge expressed as a ratio of the pre-dose baseline (SPIDnorm).

SECONDARY OUTCOMES:
Pain intensity (PI) and pain intensity difference from pre-dose baseline Time to onset of action of lozenge Assessment of redness of pharyngeal mucosa at pre-dose baseline and end of study Efficacy and tolerability assessment Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. South Africa (Pty.) Ltd.
Locations (8):
- South Africa (8):
  - Boehringer Ingelheim Investigational Site, Boksburg
  - Boehringer Ingelheim Investigational Site, Cape Town
  - Boehringer Ingelheim Investigational Site, Durban
  - Boehringer Ingelheim Investigational Site, Johannesburg
  - Boehringer Ingelheim Investigational Site, Krugersdorp
  - Boehringer Ingelheim Investigational Site, Midrand
  - Boehringer Ingelheim Investigational Site, Pretoria
  - Boehringer Ingelheim Investigational Site, Sandton